CLINICAL TRIAL: NCT05129930
Title: Fluid Overload and Pulmonary Function After Coloesophagoplasty in Children. Single-central Observational Study
Brief Title: Fluid Overload and Pulmonary Function
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: FO-Coloesopfagoplasty
Record Dates: First submitted 2021-10-07; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2020-12

CONDITIONS: Water-Electrolyte Imbalance; Intensive Care Units; Pediatric; Critical Illness; Length of Stay; Respiratory Failure; Esophageal Atresia
Keywords: Liquid; Liquid overload; Mechanical ventilation; Infant; Preschool Child; Respiratory failure; Coloesophagoplasty; Esophageal atresia
MeSH Terms: conditions — Water-Electrolyte Imbalance; Critical Illness; Respiratory Insufficiency; Esophageal Atresia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Esophageal atresia is a rare but severe malformation, and it requires early surgery. Coloesophagoplasty is surgical repair of the esophageal with an isoperistaltic transverse colon graft. In the postoperative period after coloesophagoplasty children require careful monitoring of fluid balance, because clinically significant fluid overload can lead to dysfunction of various organs and systems.

DETAILED DESCRIPTION:
Esophageal atresia (EA) is a defect of the embryogenesis of the laryngotracheal tube. There are isolated forms of EA and combinations with a tracheoesophageal fistula (TPF). Esophageal plastic surgery with an isoperistaltic transplant from the transverse colon was performed in children with EA. After this surgical intervention children require observation in the intensive care unit (ICU). During this period, infusion therapy satisfies physiological needs and compensates for physiological and pathological losses. However, it is not always possible to compensate for the body's fluid needs and maintain a normovolemic state. Thus, fluid overload develops. It is based on a pathophysiological process when severe operational stress leads to the damage of glycocalyx in the vascular wall. As a result, albumin freely passes into the interstitium, and oncotic pressure rises in tissues. Fluid overload in the intra- and postoperative period can be a factor in an unfavorable outcome, leading to organ damage, as well as death.

ELIGIBILITY:
Inclusion Criteria:

* Аge from 1 month to 3 years
* EA with / without
* Tracheoesophageal fistula (TPF)
* Сoloesophagoplasty.

Exclusion Criteria:

* Аesophageal burn,
* Oesophageal peptic stenosis,
* Congenital heart disease
* Cardiotonic support in the postoperative period
* Renal malformations
* Bacterial pneumonia in the postoperative period,
* Bronchopulmonary malformations.

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 40 children with EA with/without TPF, aged from 1 month to 3 years, who underwent coloesophagoplasty at the N.F. Filatov Children city Hospital, Moscow, Russia, from December 1, 2017 to December 31, 2020.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
duration of intensive care unit (ICU) stay | up to 30 days after the surgery
  number of days in ICU after surgery before discharge
duration of mechanical ventilation (MV) | up to 30 days after the surgery
  number of days of MV after surgery before switching to continuous positive airway pressure (CPAP)
intraoperative fluid overload (IVF) | during the surgery
  ((injected fluid (ml) - diuresis (ml) - blood loss (ml))/weight before surgery)*100%
fluid overload (FO) on the first postoperative day in the ICU | during the first postoperative day, exclude intraoperative period
  ((injected fluid (ml)-lost fluid (ml))/weight before admission to ICU)*100%
total fluid overload on the first postoperative day | during the first postoperative day, include intraoperative period
  ((injected fluid (ml) - lost fluid (ml))/weight before surgery)*100%
Fraction of Inspired Oxygen (FiO2) | in the the first postoperative day
  Fraction of Inspired Oxygen (FiO2)
Fraction of Inspired Oxygen (FiO2) | in the second postoperative day
  Fraction of Inspired Oxygen (FiO2)
Fraction of Inspired Oxygen (FiO2) | in the third postoperative day
  Fraction of Inspired Oxygen (FiO2)
Oxygen saturation (Sp02) | in the first postoperative day
  Oxygen saturation (Sp02)
Oxygen saturation (Sp02) | in the second postoperative day
  Oxygen saturation (Sp02)
Oxygen saturation (Sp02) | in the third postoperative day
  Oxygen saturation (Sp02)
Venous oxygen saturation (Svo2) | in the first postoperative day
  Venous oxygen saturation (Svo2)
Venous oxygen saturation (Svo2) | in the second postoperative day
  Venous oxygen saturation (Svo2)
Venous oxygen saturation (Svo2) | in the third postoperative day
  Venous oxygen saturation (Svo2)
partial pressure of carbon dioxide (pC02) | in the first postoperative day
  partial pressure of carbon dioxide (pC02)
partial pressure of carbon dioxide (pC02) | in the second postoperative day
  partial pressure of carbon dioxide (pC02)
partial pressure of carbon dioxide (pC02) | in the third postoperative day
  partial pressure of carbon dioxide (pC02)
inspiratory pressure (Pin) | in the first postoperative day
  inspiratory pressure (Pin)
inspiratory pressure (Pin) | in the second postoperative day
  inspiratory pressure (Pin)
inspiratory pressure (Pin) | in the third postoperative day
  inspiratory pressure (Pin)
Positive end-expiratory pressure (PEEP) | in the first postoperative day
  Positive end-expiratory pressure (PEEP)
Positive end-expiratory pressure (PEEP) | in the second postoperative day
  Positive end-expiratory pressure (PEEP)
Positive end-expiratory pressure (PEEP) | in the third postoperative day
  Positive end-expiratory pressure (PEEP)
duration of ICU stay corrected to sedation | up to 30 days after the surgery
  duration of ICU stay corrected for the duration of sedation
duration of MV corrected to sedation | up to 30 days after the surgery
  duration of MV corrected for the duration of sedation

CONTACTS AND LOCATIONS:
Overall Officials: Sergey M Stepanenko, PhD, Prof., Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- N.F. Filatov Childrens city hospital, Moscow, Russia